CLINICAL TRIAL: NCT00701610
Title: Levels of Von Willebrand Factor Multimers and VWF-Cleaving Protease (ADAMTS-13) in Preterm and Neonate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Tzipora Strauss, Sheba Medical Center
Other Study IDs: SHEBA-08-4132-TS-CTIL
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2007-07

CONDITIONS: Von Willebramd Factor
Keywords: Von Willebramd Factor (VWF); All infants born in our hospital since August 2007 ill august 2009 will enter.; Therombocytopenia, maternal aspirin will be excluded

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood will be taken from cord blood at birth from fullterm and preterm infantsinfants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All infants born in our hospital between August 2007 and August 2009 will participate.

SUMMARY:
Von Willebramd Factor (VWF) is an adhesive glycoprotein synthesized by megakaryocytes and endothelial cells.VWF has a central role in primary hemostasis and is a critical ligand for platelets adhesion and aggregation (1, 2).VWF is the carrier of circulating factor 8 as well. VWF is stored in Wiebel-Palade bodies in endothelial cells and in platelets alfa granules in a form of Ultra-large (UL) multimers.

The VWF multimers are composed from subunits which are linked by disulfide bonds that alternate between 2 C- terminal ends and 2 N- terminal ends in a head-to-head and tail-to-tail fashion (3, 4). The biological activity of VWF has been shown to be related to the size of the multimers.

VWF is released from endothelial cells toward the plasma as a multimers ranging from 500-20,000 kD. The UL multimers are hemostaticallly more effective than the smaller forms. They spontaneously bind to platelets which lead to the formation of microthrombi in the circulation. This mechanism is downregulated by the plasma protease ADAMTS-13(A Disintegrin And Metalloprotease with ThromboSpondin motif).If the proteolysis become defective the ULVWF will bind to platlets resulting in systemic thrombotic microangiophaties (TMA) such as thrombotic thrombocytopenic purpura(TTP)(5,6).

ADAMTS-13 belongs to the ADAMTS family of metalloproteases.The structure of ADAMTS-13 is conserved throughout vertebrates, indicating its important function (7).The metalloprotease function was first describe 11 years ago and has been cloned and characterized (8-13).The ADAMTS family of metaloploproteases is required in other systems such as genitourinary system (ADAMTS1), collagen system (ADAMTS2) and as a cleaving protease of VWF (VWFCP) - ADAMTS13. When VWF multimer is subjected to sufficient fluid shear stress ADAMTS-13 cleaves VWF at a unique 842Tyr- 843Met bond in domain A2 (14,15).This cleavage produce VWF subunit fragments of 176 kDa and 140 kDa.

The activity of ADAMTS-13 depends on both Zn+2 and Ca+2 ions (16). Low levels or deficiency of ADAMTS-13 is seen in patient with TTP(17,18). Mannuccio et al (19) showed that low levels of ADAMTS-13 are seen in other conditions such as healthy adults older than 65 years, patients with cirrhosis, uremia, acute inflammation, postoperative period. In neonate and preterm infants the data is limited. Few studies have shown that levels of ADAMTS-13 are low in neonate (19-21).Tsai et al (22) observed that ADAMTS-13 activity is normal in cord blood compared to adults. In preterm infants a pilot study showed that preterm have low levels of ADAMTS-13(23).

The aim of our study is to check ADAMTS-13, VWF multimers, VWF antigen and VWF collagen binding activity in healthy and sick neonate and in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* All infants born n our hospital between August 2007 and August 2009 will enter

Exclusion Criteria:

* Thrombocytopenia, maternal aspirin

Ages: 24 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants born n our hospital between August 2007 and August 2009 will enter
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Estimated); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba-Medical-Center, Ramat Gan, Israel